CLINICAL TRIAL: NCT00723502
Title: An Open-Label, Randomized, Multicenter, Two-Arms Efficacy and Safety Study of 14 Days Treatment With Finafloxacin 400 mg b.i.d. Plus Amoxicillin 1000 mg b.i.d.Versus Finafloxacin 400 mg b.i.d. Plus Esomeprazole 40 mg b.i.d. in Patients With Helicobacter Pylori Infection
Brief Title: Efficacy and Safety Study of Finafloxacin Used in Helicobacter Pylori Infected Patients
Acronym: FLASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MerLion Pharmaceuticals GmbH (Industry)
Responsible Party: Prof. Dr. P. Malfertheiner, Director, Hospiltal for Gastroenterology and Hepatology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FINA-002
Record Dates: First submitted 2008-07-25; First posted 2008-07-28 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2008-10

CONDITIONS: Gram-Negative Bacterial Infections; Helicobacter Infections; Dyspepsia
Keywords: Helicobacter pylori; Eradication; Dyspepsia
MeSH Terms: conditions — Gram-Negative Bacterial Infections; Helicobacter Infections; Dyspepsia | interventions — finafloxacin; Amoxicillin; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Finafloxacin + Amoxicillin
- 2 (Experimental)
  Interventions: Drug: Finafloxacin + Esomeprazole

INTERVENTIONS:
Drug: Finafloxacin + Amoxicillin — Finafloxacin, tablets, 400 mg b.i.d. (8 X 50 mg tablets), oral administration; Amoxicillin, tablet 1000 mg b.i.d. (1 X 1000 mg tablet), oral administration
  Arms: 1
Drug: Finafloxacin + Esomeprazole — Finafloxacin, tablets, 400 mg b.i.d. (8 X 50 mg tablets), oral administration; Esomeprazole, tablet, 40 mg b.i.d. (1 X 40 mg tablet), oral administration
  Other Names: Not apllicable
  Arms: 2

SUMMARY:
The primary objective of this study is to compare the H. pylori eradication rates with Finafloxacin in combination with Amoxicillin or Esomeprazole.

The secondary objective is to evaluate and compare the safety and tolerability of multiple oral doses of Finafloxacin plus Amoxicillin versus Finafloxacin plus Esomeprazole.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of 18 to 70 years old, with dyspepsia or dyspeptic symptoms.
2. The patient must understand the nature of the study and must provide written informed consent.
3. Each patient must be able to communicate with study personnel.
4. Gastroscopic confirmation of H. pylori infection by Rapid Urease Test.
5. Positive Urea Breath Test.
6. Absence of blood in stools.

Exclusion Criteria:

1. Gastroscopic confirmation of gastric ulcers.
2. History of Zollinger-Ellison syndrome.
3. Gastroesophageal Reflux Disease (GERD).
4. Subtotal gastrectomy or vagotomy in medical history.
5. Pyloric stenosis.
6. Previous H. pylori eradication therapy.
7. Patients likely to need to take one of the following medication within two weeks prior to and during the study period:

   * any other antibiotic than the study medication;
   * any other proton-pump inhibitor than the study medication;
   * NSAIDs including aspirin and glucocorticoids;
8. Patients taking antacids and/or H2-blockers during the study period.
9. Patients taking bismuth compound within four weeks prior to and during the study period.
10. Patients with psychiatric, neurological, or behavioral disorders that may interfere with the conduct or interpretation of the study.
11. Patients with severe concomitant disease of the cardiovascular, pulmonic, hepatic, renal, hematological, lymphatic, metabolic, and endocrine system.
12. Clinically significant serious unstable physical illness: treated, controlled and thus stable hypertension is not considered an exclusion criterion.
13. Patients with known uncontrolled hypertension or symptomatic hypotension.
14. Patients who are immunocompromised.
15. Patients with malignant disease of any kind except Basalioma.
16. Patients showing clinically significant abnormal vital signs.
17. Patients with clinically significant abnormal ECG findings.
18. Clinically significant abnormal laboratory data at Screening, or any abnormal laboratory value that could interfere with the assessment of safety.
19. Exposure to any investigational drug within 30 days prior Screening.
20. Known hypersensitivity or contraindication to the use of fluoroquinolones.
21. Prior participation in Finafloxacin study.
22. Pregnant or nursing woman, or woman of childbearing potential who is not using an effective contraceptive method during the study, e.g. oral (stable doses for at least three months prior to Screening) or injectable (stable doses for at least two months prior to Screening) contraceptives, implantation of levonorgestrel system and intrauterine devices (for at least two months prior Screening), barrier methods (combination of diaphragm and spermicide or condom and spermicide).
23. Current diagnosis or known history of substance abuse.
24. Site personnel and their immediate families, defined as their spouse, parent, child, grandparent, or grandchild.
25. Reasonable likelihood for non-compliance with the protocol or any other reason that, in the investigator's opinion, prohibits the inclusion of the patient into the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Eradication of Helicobacter pylori | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Malfertheiner, MD, Director, Principal Investigator — Not affiliated
Locations (1):
- Dr. Hein, Marburg, Germany